CLINICAL TRIAL: NCT01220713
Title: Hyperbaric Oxygen Therapy (HBO2T) for Post-Concussive Symptoms (PSC) After Mild Traumatic Brain Injury (mTBI): A Randomized, Double-Blinded, Sham Controlled, Variable Dose, Prospective Trial
Brief Title: Hyperbaric Oxygen Therapy (HBO2T) for Post-Concussive Symptoms (PSC) After Mild Traumatic Brain Injury (mTBI)
Acronym: HBOT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: United States Naval Medical Center, Portsmouth (U.S. Federal Agency); Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: N66001-09-2-2060; 01609 (Other: Hunter Holmes McGuire Veterans' Affairs Medical Center); NOMI.2010.002 (Other: Naval Operational Medical Institute); HM12204 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2010-10-06; First posted 2010-10-14 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Mild Traumatic Brain Injury; Post-Concussive Syndrome
Keywords: Traumatic Brain Injury; Veterans; Hyperbaric Oxygen Treatment; OEF/OIF; Post-Concussive Symptoms; Blast Exposure
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Brain Injuries, Traumatic | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment 1--1.5 atm abs (Experimental)
  Interventions: Procedure: Hyperbaric Oxygen Therapy
- Treatment 2--2.0 atm abs (Experimental)
  Interventions: Procedure: Hyperbaric Oxygen Therapy
- Placebo--equivalent to breathing air (Sham Comparator)
  Interventions: Procedure: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy — 1.5 atm abs oxygen equivalent of 75% oxygen (balance 25% nitrogen), 40 treatments of 60 minutes each during a time period of up to ten weeks.
  Arms: Treatment 1--1.5 atm abs
Procedure: Hyperbaric Oxygen Therapy — 2.0 atm abs oxygen equivalent of 100% oxygen (no nitrogen), 40 treatments of 60 minutes each during a time period of up to ten weeks.
  Arms: Treatment 2--2.0 atm abs
Procedure: Hyperbaric Oxygen Therapy — sham--air equivalent of 10.5% oxygen (balance 89.5% nitrogen), 40 treatments of 60 minutes each during a time period of up to ten weeks.
  Arms: Placebo--equivalent to breathing air

SUMMARY:
The goal of this research is to serve as a demonstration project to determine the tolerability of individuals with persistent post-concussive symptoms from combat-related mild TBI (traumatic brain injury), identify dose-finding for HBO2 (Hyperbaric Oxygen) therapy, and determine the efficacy of HBO2 therapy.

DETAILED DESCRIPTION:
Persistent post-concussive symptoms from mild traumatic brain injury are a severe issue facing the readiness, retention and quality of life of Department of Defense(DoD) service members and Veterans. The inadequacy of established treatment regimens and evidence-based science in post-concussive symptoms (PCS)/MTBI is forcing a closer look at non-conventional treatments of this condition. Hyperbaric oxygen (HBO2) is a potent intervention with demonstrated efficacy in dive-related injuries, soft tissue healing, and carbon monoxide poisoning.

This study is prospective, randomized, double-blinded and controlled. A total of 60 subjects will be randomly assigned to one of three treatment arms of the study: 20 subjects into the 1.5 atm abs oxygen equivalent HBO2 treatment, 20 subjects into the 2.0 atm abs oxygen equivalent HBO2 treatment and 20 subjects into the sham treatment (a placebo exposure equivalent to breathing atmospheric air). The protocol utilizes a pre- and post-treatment comprehensive performance battery that will allow for meaningful clinical outcomes and a broad understanding of the effects of the treatment. This project represents a collaboration between the Department of Defense (DoD), the Richmond Veterans Administration Medical Center (VAMC) and Virginia Commonwealth University. Service members will be recruited from military bases/treatment facilities (MTF), receive hyperbaric oxygen at existing DoD hyperbaric chambers and be evaluated by the established Virginia Commonwealth University-Center for Rehabilitation Sciences and Engineering (CERSE), a collaborative research center co-located at the Richmond VAMC and VCU.

ELIGIBILITY:
Inclusion Criteria:

1. Post-Deployment status after having served in OIF/OEF
2. Blast Event within past 3 years during OIF/OEF deployment [event defined as any of the following symptoms or experiences occurring during or shortly after the blast or explosion: dazed, confused, saw stars, headache, dizziness, irritability, memory gap (not remembering injury or injury period), hearing loss, abdominal pain, shortness of breath, struck by debris, knocked over or down, knocked into or against something, helmet damaged, evacuated]
3. Diagnosis of MTBI within 3 years as confirmed by the TBI specialty team at the Richmond VAMC
4. Presence of post-concussive symptoms from MTBI, confirmed by the VCU-CERSE team at the Richmond VAMC, for at least 3 months
5. Medical clearance to undergo hyperbaric oxygen treatment
6. Stable mental status for at least one month
7. Stable psychotropic medication history for at least one month
8. Ability to perform neuropsychologic testing battery
9. Ability to tolerate neurophysiological and neuroimaging battery

Exclusion Criteria:

1. Traumatic Brain Injury with a primary etiology other than blast
2. Moderate or Severe TBI (moderate or severe brain injury defined as best Glasgow Coma Score in first 24 hours < 12, , brain bleeding or blood clot (i.e., abnormal brain CT scan), or none of first week after event can be remembered.)
3. Past history of moderate or severe TBI
4. Active diagnosis of Post-traumatic Stress Disorder
5. Active diagnosis of Generalized Anxiety Disorder
6. Active Psychosis
7. Past history of Schizophrenia
8. Pre-existing PCS
9. Previous hyperbaric oxygen treatments
10. Contraindications to HBO2, including any "air trapping" pulmonary problems, inability to equalize middle ear and sinuses, or patients who are claustrophobic and require anti-anxiety medication for the condition
11. Active use of cancer medications
12. Pregnancy

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Improvement on symptom assessment battery | 2-4 weeks before treatment
  Symptom Assessment Battery include: Rivermead Postconcussive Symptom Questionnaire, Pain Intensity Numerical 0-10 scale, Alcohol Use Disorders Test-Consumption, McGill Pain Questionnaire-Short Form, The Center for Epidemiological Studies Depression Scale, PTSD Checklist-Military Version, Extended Glasgow Outcome Scale, Mayo-Portland Adaptability Inventory 4, Satisfaction With Life Scale
Improvement on symptom assessment battery | 24-72 hours after final treatment
  Symptom Assessment Battery include: Rivermead Postconcussive Symptom Questionnaire, Pain Intensity Numerical 0-10 scale, Alcohol Use Disorders Test-Consumption, McGill Pain Questionnaire-Short Form, The Center for Epidemiological Studies Depression Scale, PTSD Checklist-Military Version, Extended Glasgow Outcome Scale, Mayo-Portland Adaptability Inventory 4, Satisfaction With Life Scale
Improvement on symptom assessment battery | 3 months after final treatment.
  Symptom Assessment Battery include: Rivermead Postconcussive Symptom Questionnaire, Pain Intensity Numerical 0-10 scale, Alcohol Use Disorders Test-Consumption, McGill Pain Questionnaire-Short Form, The Center for Epidemiological Studies Depression Scale, PTSD Checklist-Military Version, Extended Glasgow Outcome Scale, Mayo-Portland Adaptability Inventory 4, Satisfaction With Life Scale

SECONDARY OUTCOMES:
Neuropsychological Testing Battery | 2-4 weeks before treatment
  Test Battery Includes: Trail Making Test, Stroop Classic, California Verbal Learning Test-II, Wechsler Test of Adult Reading, Wechsler Adult Intelligence Scale III (WAIS-III): Digit Symbol Coding Digit Span Letter-Number Sequencing Symbol Search and Arithmetic, Delis-Kaplan Executive Functioning System(D-KEFS): Controlled Oral Word Exam (COWA), Grooved Pedboard, Test of Memory Malingering, Benton Visual Memory Test-Revised
Neurophysiologic Measures of Human Performance: Computerized Posturography, NeuroImaging and Eye tracking | 24-72 hours after final treatment
Common Military Task Tests | 2-4 weeks before treatment
  Testing includes: Mission-oriented protective posture (MOPP) gear donning, Protective mask usage, personal weapon assembly/dis-assembly, grenade inspection/identification, acute management of injury-induced shock
Neuropsychological Testing Battery | 24-72 hours after final treatment
  Test Battery Includes: Trail Making Test, Stroop Classic, California Verbal Learning Test-II, Wechsler Test of Adult Reading, Wechsler Adult Intelligence Scale III (WAIS-III): Digit Symbol Coding Digit Span Letter-Number Sequencing Symbol Search and Arithmetic, Delis-Kaplan Executive Functioning System(D-KEFS): Controlled Oral Word Exam (COWA), Grooved Pedboard, Test of Memory Malingering, Benton Visual Memory Test-Revised
Neurophysiologic Measures of Human Performance: Computerized Posturography, NeuroImaging, Eye tracking | 3 months after final treatment.
Neuropsychological Testing Battery | 3 months after final treatment.
  Test Battery Includes: Trail Making Test, Stroop Classic, California Verbal Learning Test-II, Wechsler Test of Adult Reading, Wechsler Adult Intelligence Scale III (WAIS-III): Digit Symbol Coding Digit Span Letter-Number Sequencing Symbol Search and Arithmetic, Delis-Kaplan Executive Functioning System(D-KEFS): Controlled Oral Word Exam (COWA), Grooved Pedboard, Test of Memory Malingering, Benton Visual Memory Test-Revised
Neurophysiologic Measures of Human Performance: Computerized Posturography, NeuroImaging, Eye tracking | 2-4 weeks before treatment
Common Military Task Tests | 24-72 hours after final treatment
  Testing includes: Mission-oriented protective posture (MOPP) gear donning, Protective mask usage, personal weapon assembly/dis-assembly, grenade inspection/identification, acute management of injury-induced shock
Common Military Task Tests | 3 months after final treatment.
  Testing includes: Mission-oriented protective posture (MOPP) gear donning, Protective mask usage, personal weapon assembly/dis-assembly, grenade inspection/identification, acute management of injury-induced shock

CONTACTS AND LOCATIONS:
Overall Officials: David X Cifu, MD, Principal Investigator — Virginia Commonwealth University; Brett Hart, MD, Principal Investigator — Naval Operational Medicine Institute; Michelle Nichols, MSN, RN, Principal Investigator — McGuire Veterans' Affairs Medical Center; Justin O Alicea, Study Director — Virginia Commonwealth University; Steven L West, PhD, Study Director — Virginia Commonwealth University
Locations (3):
- United States (3):
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - Hunter Holmes McGuire Veterans' Affairs Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia